CLINICAL TRIAL: NCT03975608
Title: Adaptation of a Psychological Therapy for Patients With ALS - a Pilot Study
Brief Title: Psychological Therapy for Patients With ALS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Anja Mehnert, Head of the Department of Medical Psychology and Medical Sociology, University of Leipzig
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ALS_Pilot
Record Dates: First submitted 2019-05-23; First posted 2019-06-05 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Amyotrophic Lateral Sclerosis; Psychological Stress
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Stress, Psychological

STUDY DESIGN:
Intervention Model Description: The design of this project will be a non-randomised and non-controlled before-and-after study in which observations will be made only in a patient group that receives the intervention. No control group will be recruited. Assessments will be conducted at three measurement points: T0 (before the intervention), T1 (at the end of the intervention), T2 (3 months after T1).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adaptation of "CALM" (Experimental): This is the patient group that receives the intervention (IG), i.e., the psychotherapeutic treatment, i.e., the adapted version of the psychotherapeutic program "Managing Cancer and Living Meaningfully (CALM)" which was originally designed for patients with cancer.
  Interventions: Behavioral: Adaptation of "CALM"

INTERVENTIONS:
Behavioral: Adaptation of "CALM" — The therapy is built up by 3-8 sessions (duration about 45-60 min) over a period of 6 months. All dimensions are explored with every patient, but the order and extent of each dimension are adapted to the individual needs of the patient.
  The sessions address the 4 dimensions of the original program designed for palliative cancer patients:
  1. Symptom management and communication with healthcare providers
  2. Changes in self and relations with each others
  3. Spirituality, sense of meaning, and purpose
  4. Thinking of the future, hope, and mortality
  As an adaptation, the investigators will especially focus on two other aspects which take into account the specific symptoms and challenges in patients with ALS: (i) communication skills and (ii) emotional expression and control.

SUMMARY:
Amyotrophic lateral sclerosis (ALS) is a disease that is inevitably fatal. To be diagnosed with a terminal illness such as ALS deeply affects one's personal existence and goes along with significant changes regarding the physical, emotional, and social domains of the patients' life. This pilot study will test a manualized, individual psychotherapeutic intervention to relieve distress and promote psychological well-being in ALS patients. A total of 5 patients will receive the intervention. The investigators will gather important information regarding the feasibility of the intervention (i.e., response rate, patient and therapist adherence, and patient satisfaction), which may be used for conducting a future randomized controlled trial. Various domains of quality of life will be assessed before the intervention (T0), after the intervention (T1) and at 3-months-follow-up (T2) in order to test for preliminary efficacy of the intervention.

DETAILED DESCRIPTION:
Background: Amyotrophic lateral sclerosis (ALS) is a progressive neurodegenerative disease that is inevitably fatal. To be diagnosed with a terminal illness such as ALS deeply affects one's personal existence and goes along with significant changes regarding the physical, emotional, and social domains of the patients' life. ALS patients have to face a rapidly debilitating physical decline which restrains mobility and impairs all activities of daily living. In addition, they are confronted with their own mortality. This progressive loss of autonomy and fears about the future may lead to a sense of hopelessness and loss of quality of life, which in turn may even result in thoughts about physician-assisted suicide.

Concrete aims: Given the high emotional strain in this patient group, this study aims to apply a manualized psychotherapeutic intervention to relieve distress and promote psychological well-being on ALS patients. This short-term intervention (up to six sessions) was originally developed for advanced cancer patients. "Managing Cancer and Living Meaningfully (CALM)" focuses on the four dimensions: (i) symptom management and communication with healthcare providers, (ii) changes in self and relations with close others, (iii) spirituality, sense of meaning and purpose and (iv) thinking of the future, hope, and mortality.

Methodology: For these aims mentioned above, the investigators will conduct a feasibility study, i.e., a pilot study before a future randomized controlled trial can be planned in detail. The design of this pilot intervention will be a non-randomised prospective non-controlled before-and-after study, in which observations will be made only in a patient group (n = 5) that receives the intervention (IG). No control group will be recruited. Assessments will be conducted on the three measurement points: before the therapy (T0), after the intervention (T1) and 3 months after the intervention (T2).This study is intended to test out the standard operating procedures, evaluate the feasibility, acceptance and adherence to the study protocol as well as preliminary efficacy of the intervention.

Recruitment: Patients will be consecutively recruited in the Clinic of Neurology at the University Medical Center of Leipzig.

Duration: The duration for patients will be about 9 months (6 months intervention, 3 month-follow-up assessment). The duration of the whole study will be 12 months.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of Amyotrophic Lateral Sclerosis
* minimum age of 18 years
* fluent in German language
* ability to visit the institution providing the intervention at the start of therapy (in the course of treatment, telephone-sessions may be offered)
* ability to report on thoughts and feelings (by speaking, writing or via communication devices)
* cognitive ability to give written informed consent
* expected remaining lifetime of at least 9 months

Exclusion Criteria:

* inability for communicate (neither via speaking, writing or communication devices)
* currently in psychotherapeutic treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-11-15 (Actual)

PRIMARY OUTCOMES:
Response rate | The assessment period for this outcome will be from the start of recruitment until the inclusion of the last patient, which will be about 1 year.
  The investigators will assess the amount of eligible patients which are willing to participate in the study relative to the amount of patients who were invited to participate.
Patient adherence | During the intervention phase for each patient, which will be about sixth months.
  Patient adherence will be assessed via documentation of patient drop-outs. In detail, we will document whether patients leave the study during the treatment (and if yes, at what stage).
Patient satisfaction | Assessed only once for each patient, immediately after the patient has completed the intervention.
  Assessed by a questionnaire (Working Alliance Inventory - short form revised). The total sum score across the 12 items, rated on a five-point Likert scale, will be presented (ranging from 12 to 60). Higher values present higher satisfaction.

SECONDARY OUTCOMES:
Level of quality of life | Assessed at three time points: before the intervention, immediately after the intervention and 3 months after the intervention
  Assessed by a questionnaire, the Amyotrophic Lateral Sclerosis Assessment Questionnaires - short form (ALSAQ-5). The total score across the 5 items, rated on a 4-point Likert scale, will be presented (range: 0 - 20). Higher values indicate higher quality of life.
Level of depressive symptomatology | Assessed at three time points: before the intervention, immediately after the intervention and 3 months after the intervention
  Assessed by a questionnaire, the ALS-Depression-Inventory (ADI-12). The sum score across all 12 items, each rated on a 4-point Likert-scale, will be reported (range: 12-48). Higher values indicate higher levels of depression.
Level of functioning | Assessed at three time points: before the intervention, immediately after the intervention and 3 months after the intervention
  Assessed by a questionnaire, the revised Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS-R). The total sum score across the 15 items, each rated on a 5-point LIkert scale, will be reported (range: 0-60). Higher values indicate a higher level of functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Anja Mehnert-Theuerkauf, Prof. Dr., Principal Investigator — University of Leipzig; Joseph Claßen, Prof. Dr., Principal Investigator — University of Leipzig
Locations (1):
- University Medical Center Leipzig, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Metelmann M, Heyne S, Peuker M, Classen J, Mehnert-Theuerkauf A, Esser P. [Experiences with the Application of Short-Term Psychotherapy in Patients with Amyotrophic Lateral Sclerosis: What Can We Learn from It?]. Psychother Psychosom Med Psychol. 2025 Nov 12. doi: 10.1055/a-2711-2085. Online ahead of print. German. PMID 41224202